CLINICAL TRIAL: NCT05533489
Title: Risk Factors for Postoperative Pain After Arthroscopic Anterior Cruciate Ligament Reconstruction
Brief Title: Risk Factors for Post ACL Reconstruction Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Sasikaan Nimmaanrat, Associate Professor, Prince of Songkla University
Other Study IDs: REC.65-319-8-1
Record Dates: First submitted 2022-09-05; First posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Risk Factors for Post ACL Reconstruction Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention This study is a retrospective descriptive study.

SUMMARY:
In 2006, approximately 130,000 arthroscopic anterior cruciate ligament reconstructions were performed in the United States, and the number is increasing each year. Despite being a minimally invasive procedure, pain is the most common postoperative problem after arthroscopic anterior cruciate ligament reconstruction associated with cost, postoperative opioid consumption, opioid-related side effects, quality of life, patient satisfaction, and delayed discharge. Over two-thirds of the patient receiving arthroscopic anterior cruciate ligament surgery have moderate to severe pain.

DETAILED DESCRIPTION:
At present, multimodal analgesia is a successful mainstay treatment for arthroscopic anterior cruciate ligament surgery which range from opioid, paracetamol, non-steroidal anti-inflammatory agents (NSAIDs), local anesthetic agents, ketamine, corticosteroid, and cold compression therapy. Previous study showed femoral nerve block reduces pain score but also increases incidence of falling. Afterward, a study on adductor canal block showed equivalent postoperative analgesia while preserving quadriceps strength. Furthermore, a few studies were conducted to determine risk factors for postoperative pain after arthroscopic anterior cruciate ligament surgery, but results are contradictory. Previous research found risk factors for postoperative pain after arthroscopic anterior cruciate ligament surgery are female, young age, smoker, preoperative visual analog scale score ≥3, tourniquet time > 50 minutes, and cartilage injury. In addition, evidence showed higher preoperative visual analog scale, and previous opioid use are associated with greater amount of opioid consumption. In contrary, some evidence showed no effect of age, sex, body mass index (BMI), tourniquet time, type of anesthesia on post postoperative pain after arthroscopic anterior cruciate ligament surgery.

ELIGIBILITY:
Patients undergoing primary unilateral arthroscopic anterior cruciate ligament reconstruction with or without unilateral cartilage/meniscus injury with or without other ligaments injury (posterior cruciate ligament/medial collateral ligament/lateral collateral ligament) Age ≥ 15 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary unilateral arthroscopic anterior cruciate ligament reconstruction with or without unilateral cartilage/meniscus injury with or without other ligaments injury (posterior cruciate ligament/medial collateral ligament/lateral collateral ligament)
Sampling Method: Non-Probability Sample
Enrollment: 924 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To find risk factors for moderate to severe postoperative pain after arthroscopic anterior cruciate ligament reconstruction in the first 72 hours. | Three days
  To find risk factors for moderate to severe postoperative pain after arthroscopic anterior cruciate ligament reconstruction in the first 72 hours

SECONDARY OUTCOMES:
To find incidence of moderate to severe pain after arthroscopic anterior cruciate ligament reconstruction in the first 72 hours | Three days
  To find incidence of moderate to severe pain after arthroscopic anterior cruciate ligament reconstruction in the first 72 hours
To find analgesic requirement after arthroscopic anterior cruciate ligament reconstruction for 1 year | One year after discharge
  To find analgesic requirement after arthroscopic anterior cruciate ligament reconstruction for 1 year

IPD SHARING:
Plan to Share IPD: Undecided